CLINICAL TRIAL: NCT05909826
Title: A Phase II Study of Carfilzomib, Oral Cyclophosphamide, and Dexamethasone for Relapsed and/or Refractory Multiple Myeloma
Brief Title: Carfilzomib, Oral Cyclophosphamide, and Dexamethasone for RRMM
Acronym: KMM-KCd
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Hyun Kim, Professor, Dong-A University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAUHIRB-23-038
Record Dates: First submitted 2023-02-28; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Weekly carfilzomib-oral cyclophosphamide-dexamethasone (Experimental): Weekly carfilzomib-oral cyclophosphamide-dexamethasone
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — 70 mg/m2 IV days 1, 8 and 15, every 4 weeks
  Other Names: Kyprolis
Drug: Cyclophosphamide — 50 mg PO days 1 to 21, every 4 weeks
  Other Names: Alkyloxan
Drug: Dexamethasone — 40mg PO or IV days 1, 8, 15, and 22, every 4 weeks

SUMMARY:
This study aims to study the efficacy and safety of oral cyclophosphamide in addition to carfilzomib and dexamethadone for RRMM patients who have been previously exposed to lenalidomide combination therapies.

DETAILED DESCRIPTION:
The survival of multiple myeloma (MM) patients has been improved significantly owing to the adoption of immunomodulatory agents (IMiD) and proteasome inhibitors (PI). However, most of the MM patients finally experience relapse of refractoriness of the disease, of which patients who relapse after bortezomib and lenalidomide have very poor prognosis. Carfilzomib is an irreversible second generation PI which is approved by Korean FDA for RRMM in combination with dexamethasone and/or lenalidomide based on the landmark studies ASPIRE and ENDEAVOR studies. The addition of intravenous cyclophosphamide to carfilzomib has recently showed a promising result for RRMM patients after bortezomib and lenalidomide. In this study, cyclophosphamide 50mg orally will be added to carfilzomib once weekly schedule for 21 days daily every 4 weeks. The rationale for oral metronomic cyclophosphamide is based on previous experimental studies which has shown that it removes CD4+CD25+regulatory T cells preserving T and NK/T cell funtions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 19 years or older
2. ECOG performance status 0 to 2
3. Diagnosed with multiple myeloma by IMWG criteria
4. Subjects previously treated with 1 or more lines of therapy
5. Subjects previously treated with lenalidomide-based combination or sigle drug therapy
6. Subjects with relapsed and/or refractory multiple myeloma
7. Subjects with measurable disease at the time of treatment initiation

   * serum M protein >=0.5 g/dL, or
   * 24h urine M protein >= 200mg/24h
   * serum free light chain difference >=10mg/dL and abnormal FLC ratio
8. Adequate organ function

   * absolute neutrophil count >= 1.0 x 109/L
   * platelelt count >= 50 x 109/L (plasmacytoma in the bone: >=30 x 109/L)
   * Hb >=8g/dL
   * serum creatinine < 3.0mg/dL or CCR >=15mL/min
   * serum AST and ALT <=3 x ULN
   * serum total bilirubin <= 3 x ULN
9. Subjects able to swallow oral drugs
10. Subjects who had experienced toxicities to previous therapies: resolved from previous toxicities or stabilized of the toxicity to grade 1
11. Subjects who had received allogenetic stem cell transplantation: no acitve graft-versus-host disease
12. Subjects without clinically relevant bleeding
13. Subjects who have informed consent to the study
14. Females of childbearing potential (FCBP) must be negative to pregnancy testing and give consent to practice contraception before and during the treatment

Exclusion Criteria:

1. Subjects who were previously exposed to carfilzomib

1. Subjects who were previously exposed to cyclophosphamide 3. Subjects diagnosed with POEMS SD, Waldenstrom macroglobulinemia, Plasma cell leukemia 4. Subjects with concurrent heart conditions

* Myocardial infarction within 6 months prior to treatment, New York Heart Association class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease,
* Uncontrolled arrythmias (CVDAE version4 grade 2 or more) or symptomatic EKG abnormalities
* 12-lead EKG : baseline ATcF > 470msec
* 2D Echocardiography or MUGA scan : systolic EF < 40% with clinically significant symptoms
* Uncontrolled hypertension ( with medication: systolic BP >= 160 mmHg or diastolic BP >= 100 mmHg) 5. Chronc obstructive pulmonary disease (FEV1 < 60%), history of asthma within 2 years 6. Surgery under general anesthesia withing 2 weeks 7. Subjects diagnosed with malignancies within 5 years (except for cured skin cancer, cervical cancer, intraepithelial gastrointestinal tract cancer after curative procedures or surgery for more than 3 years) 8. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent 9. Pregnant or breatfeeding subjecs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Very good partial response | from the first date of KCd to the day 30 after KCd stop date
  Reduction of serum M-protein > 90%

SECONDARY OUTCOMES:
Overall response | from the first date of KCd to the day 30 after KCd stop date
  sCR+CR+VGPR+PR
Progression-free survival | from the first date of KCd until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  the time from the first date of KCd to the date of disease progression or death or censored date
Overall survival | from the first date of KCd until the date of death from any cause, assessed up to 48 months
  the time from the first date of KCd to the date of death or censored date
Duration of response | from the first date of PR to the date of disease progression or death or censord date, which ever came first, assessed up to 48 months
  the time from the first date of PR to the date of disease progression or death or censord date
Time to response | from the first date of KCd to the date of first date of equal or more than partial response, which ever came first, assessed up to 48 months
  the time from the first date of KCd to the first date of partial response
Safety profile | from the first date of KCd to day 30 after KCd stop date
  Adverse events after KCd

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hyun Kim, MD, Ph.D, Principal Investigator — Dong-A University

IPD SHARING:
Plan to Share IPD: No